CLINICAL TRIAL: NCT02485080
Title: Safety, Tolerability, and Efficacy of Simeprevir 150 mg Daily Plus Sofosbuvir 400 mg Daily for 24 Weeks in Patients With Chronic Hepatitis C Genotype 1 With CPT Score of 6 or Lower Who Are IFN-Intolerant or Unwilling to be Treated With IFN
Brief Title: Safety, Tolerability, and Efficacy of 24 Weeks Simeprevir+Sofosbuvir for Chronic Hepatitis C Genotype 1
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawn due to lack of resources
Sponsor: Stanford University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Yale University (Other)
Responsible Party: Principal Investigator, Mindie H. Nguyen, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33431
Record Dates: First submitted 2015-06-23; First posted 2015-06-30 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: PT-NANBH
Keywords: hepatitis C; liver transplantation; genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simeprevir + sofosbuvir daily, 24 weeks (Experimental): Eligible and consenting patients will be treated with sofosbuvir (SOF) 400 mg daily and simeprevir (SMV) 150 mg daily for 24 weeks. Both drugs will be administered orally, per manufacturers' instructions.
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Simeprevir
  Other Names: Olysio
Drug: Sofosbuvir
  Other Names: Sovaldi

SUMMARY:
The goal of this pilot study is to examine both efficacy and tolerability in patients with HCV genotype 1 and mild decompensation with Child-Pugh-Turcott score of 6 or lower. The CPT score is used to assess the prognosis of chronic liver diseases, as well as the required strength and treatment and necessity of liver transplantation. A higher CPT score denotes higher necessity of liver transplantation.

DETAILED DESCRIPTION:
Key objectives of this study include:

1. To describe efficacy (SVR) in a special population of patients with chronic hepatitis C who are not willing or not candidates for IFN-based therapy.
2. To describe safety, tolerability, and treatment persistency in this patient population with advanced liver disease.

ELIGIBILITY:
Inclusion criteria:

1. Adult 18-72 years
2. Cirrhosis: defined by stage 4 on biopsy or noninvasive tests or presence of splenomegaly and platelet of 130K or lower, or presence of shrunken nodular liver on CT or MRI, or presence of varices or encephalopathy or ascites.
3. HCV genotype 1 or indeterminate and later assessed at Screening and confirmed as genotype 1

Exclusion criteria:

1. Uncontrolled ascites, uncontrolled hepatic encephalopathy, or uncontrolled esophageal/gastric varices
2. Co-infection with HIV or hepatitis B (HBV)
3. CPT 7 or above, or MELD >10
4. Total bilirubin 4.0 mg/dL or above
5. CrCl (creatinine clearance) < 30 mL/min
6. Any unstable active medical illnesses.
7. Active use of illicit substances, alcohol, or smoking.
8. Any malignancy within last 5 years except for basal cell skin cancer that has been adequately treated or HCC within Milan or UCSF criteria, which will be acceptable
9. Any prior treatment with direct acting antivirals (approved or investigational), including HCV protease inhibitors, such as SMV. Patients who received prior treatment with SOF, and/or NS5A inhibitors (e.g. ledipasvir or Daclatasvir) can be included in this study
10. Platelet < 30 K/uL

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) HCV RNA PCR <25 IU/mL 12 weeks post-treatment | 12 weeks after end of treatment or virologic response after liver transplantation, whichever comes first, assessed up to 12 weeks after end of treatment

SECONDARY OUTCOMES:
Serious adverse events, adverse events grade 3 and above | 24 weeks while on treatment and 24 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mindie H Nguyen, MD, MAS, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University Medical Center, Palo Alto, California
  - Yale University Medical Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roche B, Samuel D. Hepatitis C virus treatment pre- and post-liver transplantation. Liver Int. 2012 Feb;32 Suppl 1:120-8. doi: 10.1111/j.1478-3231.2011.02714.x. PMID 22212582
- [Background] Carrion JA, Martinez-Bauer E, Crespo G, Ramirez S, Perez-del-Pulgar S, Garcia-Valdecasas JC, Navasa M, Forns X. Antiviral therapy increases the risk of bacterial infections in HCV-infected cirrhotic patients awaiting liver transplantation: A retrospective study. J Hepatol. 2009 Apr;50(4):719-28. doi: 10.1016/j.jhep.2008.11.015. Epub 2008 Dec 29. PMID 19217183
- [Background] Iacobellis A, Siciliano M, Perri F, Annicchiarico BE, Leandro G, Caruso N, Accadia L, Bombardieri G, Andriulli A. Peginterferon alfa-2b and ribavirin in patients with hepatitis C virus and decompensated cirrhosis: a controlled study. J Hepatol. 2007 Feb;46(2):206-12. doi: 10.1016/j.jhep.2006.08.020. Epub 2006 Oct 20. PMID 17125876
- See also: Recommendations for Testing, Managing, and Treating Hepatitis C by the American Association for the Study of Liver Diseases and Infectious Disease Society of America — http://www.hcvguidelines.org
- See also: OLYSIO (Simeprevir) package insert — https://www.olysio.com/shared/product/olysio/prescribing-information.pdf
- See also: SOLVALDI (Sofosbuvir) package insert — https://www.gilead.com/~/media/Files/pdfs/medicines/liver-disease/sovaldi/sovaldi_pi.pdf